CLINICAL TRIAL: NCT00478036
Title: A Randomized Prospective Double Masked Controlled Trial Comparing Ketorolac Tromethamine 0.4% and Prednisolone Acetate 1% in Reducing Post-selective Laser Trabeculoplasty Anterior Chamber Flare and Cells.
Brief Title: Comparing Acular LS and Pred Forte in Reducing Post-selective Laser Trabeculoplasty Anterior Chamber Flare and Cells
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-1251
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Open Angle Glaucoma
Keywords: glaucoma; selective laser trabeculoplasty; anterior chamber flare
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Ketorolac; Ketorolac Tromethamine; Ophthalmic Solutions; prednisolone acetate; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acular LS (Active Comparator): Acular LS - 1 drop in treated eye, 4 times a day, for 4 days
  Interventions: Drug: Acular LS
- Pred Forte (Active Comparator): Pred Forte - 1 drop in treated eye, 4 times a day, for 4 days
  Interventions: Drug: Pred Forte
- Refresh Tears (Placebo Comparator): Refresh Tears - 1 drop in treated eye, 4 times a day, for 4 days
  Interventions: Other: Refresh Tears

INTERVENTIONS:
Drug: Acular LS — Details covered in arm description
  Other Names: KETOROLAC TROMETHAMINE 0.5% SOLUTION - OPHTHALMIC
  Arms: Acular LS
Drug: Pred Forte — Details covered in arm description
  Other Names: Prednisolone acetate ophthalmic suspension 1%
  Arms: Pred Forte
Other: Refresh Tears — Placebo
  Other Names: CARBOXYMETHYLCELLULOSE SODIUM
  Arms: Refresh Tears

SUMMARY:
The Investigators will compare, in a randomized, prospective, masked and controlled fashion the effect of a non-steroidal anti-inflammatory agent (Acular LS), a corticosteroid (Pred Forte) and a placebo (Refresh Tears) on patient discomfort, degree of intraocular pressure (IOP) lowering and degree of ocular inflammation following selective laser trabeculoplasty treatment for open angle glaucoma.

DETAILED DESCRIPTION:
Currently, many ophthalmologists use anti-inflammatory agents like corticosteroids and nonsteroidal anti-inflammatory agents (NSAIDs) as a preventative measure to control the post-selective laser trabeculoplasty (SLT) anterior chamber inflammation. Both classes of compounds reduce inflammation through the inhibition of the cyclooxygenase pathway, whereas the corticosteroid class also inhibits the lipoxygenase pathway of the arachidonic acid cascade. Although effective, topical corticosteroids are associated with increase in intraocular pressure (IOP), posterior subcapsular cataract formation, and reduced response to infection. These adverse side effects have not been reported to occur with topical NSAIDs, which are effective in controlling the pain after SLT along with the prevention and suppression of the ocular inflammation. There are ophthalmologists who forgo using the anti-inflammatory agents post SLT and prescribe Refresh Tears to their patients to comfort the treated eye.

The significance of the study lies in assessing the efficacy of Acular LS, compared to Pred Forte and to Refresh Tears in reducing discomfort, inflammation and maximizing IOP lowering following SLT procedure for open angle glaucoma with the hope of resolving the dispute over the effective post-operative care in SLT patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open angle glaucoma patients at the Rocky Mountain Lions Eye Institute Glaucoma Clinic.
* Able to provide written informed consent to participate.
* Must be the age of 18 years of age or older.
* Patients in which further intraocular pressure lowering by selective laser trabeculoplasty is necessary in the opinion of the treating physician.

Exclusion Criteria:

* Patients with eye surgery in the prior six months.
* Patients with prior or current use of topical or systemic corticosteroids or NSAIDs.
* Patients with pre-existing anterior chamber inflammation.
* Patients with known sensitivity to any of the study medications.
* Due to the age range and the disease entity, special patient populations such as children or pregnant women will not be enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — Rocky Mountain Lions Eye Institute
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective study participants will be identified by a routine clinic visit at Rocky Mountain Lions Eye Institute, University of Colorado, and need to undergo selective laser trabeculoplasty treatment for their glaucoma. A study investigator will make the initial patient contact for recruitment.
Pre-assignment Details: The patients enrolled in this study will follow standard of care practice in regards to selective laser trabeculoplasty with the exception that the patients will be randomized 1:1:1 (Acular LS: Pred Forte: Refresh Tears) to the inflammation treatment given after the procedure.
Period: Overall Study
Arm/Group | Acular LS | Pred Forte | Refresh Tears
Started | 10 | 7 | 14
Completed | 10 | 7 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Refresh Tears - 1 drop in treated eye, 4 times a day, for 4 days
- Acular Group: Used acular LS
- Predforte Group: Used predforte eye drops
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Acular Group | Predforte Group | Total
Number analyzed (Participants) | 14 | 10 | 7 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 1 | 8
  >=65 years | 11 | 6 | 6 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [62 to 71] | 69.5 [60.5 to 73] | 73 [66.5 to 77.5] | 69 [63 to 72.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 3 | 22
  Male | 1 | 4 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Interocular Pressure
Description: IOP, measured by Goldmann applanation tonometry
Time Frame: 8 weeks
Population: Reported for subjects for whom all IOP values were available for all of the visits.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Acular LS | Pred Forte | Refresh Tears
Number analyzed (Participants) | 9 | 7 | 11
mmHg
  Baseline | 16.1 (3.1) | 17.0 (3.3) | 17.8 (4.5)
  Day 1 | 11.6 (2.2) | 12.4 (2.5) | 13.4 (3.3)
  Week 1 | 15.2 (3.3) | 15.7 (2.8) | 15.6 (3.7)
  Week 4 | 14.3 (2.6) | 14.0 (2.4) | 14.6 (3.5)
  week 8 | 14.0 (2.3) | 15.0 (1.6) | 15.8 (3.1)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Acular LS | Pred Forte | Refresh Tears
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No